CLINICAL TRIAL: NCT04666506
Title: Relaxation-VR: Implementation of Virtual Reality for Children in Hospital
Acronym: Relaxation-VR
Status: Completed | Type: Observational
Sponsor: Thomas More University of Applied Sciences (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other); Algemeen Ziekenhuis Sint_Maarten (Unknown)
Responsible Party: Sponsor
Other Study IDs: IC_PED_01
Record Dates: First submitted 2020-12-01; First posted 2020-12-14 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Anxiety; Pain; Stress
Keywords: Virtual reality; VR; paediatric; distraction; pain; anxiety; relaxation
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VR as distraction during a medical procedure: Paediatric outpatients undergoing a medical procedure, aged 4-16 years old in Belgian hospitals UZ Brussel and AZ Sint-Maarten, will use VR as a distraction method during a potentially painful or scary procedure (e.g., vaccination, wound care, venipuncture,...).
  Interventions: Other: Virtual reality
- VR as relaxation method during a hospital stay: Paediatric inpatients, aged 4-16 years old in Belgian hospitals UZ Brussel and AZ Sint-Maarten, will use VR as a relaxation method during a potentially stressful hospital stay (e.g., patients with psychosomatic complaints, patients with eating disorders,...).
  Interventions: Other: Virtual reality

INTERVENTIONS:
Other: Virtual reality — The VR intervention, Relaxation-VR, is a VR application developed by Psylaris aiming to reduce anxiety/stress and pain by distracting the patient in a relaxing environment. Relaxation-VR will be administered via a commercially available VR headset (Oculus Go). The VR headset is a piece of equipment that a person wears over their eyes that allows them to experience images and sounds produced by a computer as if they were part of real life (Cambridge Dictionary, 2020). As such, the patient is immersed in a novel, calming and distracting environment where the he/she is asked to perform tasks that will help the patients to relax when distressed before and/or during a medical procedure or during their stay in hospital.
  The Relaxation-VR application consists of three modules: two modules make use of relaxation principles (i.e. breathing exercises, meditation) and one module presents a scene with different interactive animations and objects (i.e. popping bubbles, playing fetch with a dog).
  Other Names: Relaxation-VR

SUMMARY:
Although on an international level, accumulating evidence supports the feasibility and effectiveness of VR for pain and anxiety management, in Belgium, adoption of VR in clinical practice is limited and local trials are scarce. In order to improve translation from research to practice, the current study will focus on the feasibility, acceptability, tolerability and preliminary effectiveness of 'Relaxation-VR', a VR application aiming to reduce anxiety and pain for children admitted to hospital, as experienced by both patients and clinical staff. This study will take place at the paediatric wards of two hospitals interested in adopting this innovative technology for improving both patient care (e.g., anxiety and pain reduction) and staff workload (e.g., shorter procedure times), UZ Brussel and AZ Sint-Maarten.

DETAILED DESCRIPTION:
Current pain and anxiety management for children in hospital includes pharmacological analgesia (e.g. opioid therapy) with potential negative side effects. In addition, a non-pharmacological approach involves various distraction techniques, either passive (e.g., music, movies) or active (e.g., interactive toys, electronic games, storytelling by the nursing staff). However, these distraction techniques can often be time consuming for the already busy and even over-demanded nursing staff.

A combination of distraction, extinction learning, cognitive-behavioral principles, mindful meditation, stress reduction, gate-control theory, and the spotlight theory of attention is believed to be the mechanism behind VR's effectiveness in pain management. Accumulating evidence supports VR as a feasible and effective method to alleviate anxiety and pain for paediatric patients during lumbar punctures, intravenous injections, burn wound care and rehabilitation. In particular, a recent meta-analysis reported that the use of VR was significantly more effective in reducing pain (14 studies) and anxiety (7 studies) than care as usual (CAU), with large effect size. Moreover, for chest radiography, the use of VR has also significantly reduced procedure time, while increasing patient satisfaction. As such, adding the use of VR to standard pain and anxiety management methods might improve both effectiveness and efficiency of current practice.

Although on an international level, accumulating evidence supports the feasibility and effectiveness of VR for pain and anxiety management, in Belgium, adoption of VR in clinical practice is limited and local trials are scarce. In order to improve translation from research to practice, the current study will focus on the feasibility, acceptability, tolerability and preliminary effectiveness of 'Relaxation-VR', a VR application aiming to reduce anxiety and pain for children admitted to hospital, as experienced by both patients and clinical staff. This study will take place at the paediatric wards of two hospitals interested in adopting this innovative technology for improving both patient care (e.g., anxiety and pain reduction) and staff workload (e.g., shorter procedure times), UZ Brussel and AZ Sint-Maarten.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained
* Inpatient or outpatient in one of the study sites (UZ Brussel or AZ Sint-Maarten): each paediatric patient who will undergo treatment or a single medical (nursing) procedure during the study period (1-01-2021 and 30-09-2021) and is in need of relaxation or distraction, as assessed by the clinical expertise of the involved clinical staff*.

  * For example (but not limited to), for the relaxation module of the VR intervention, following paediatric patients can be recruited: paediatric patients awaiting surgery, paediatric patients post-surgery during their (brief) stay in the recovery unit, paediatric patients staying at the oncological department, paediatric patients with eating disorders in need of relaxation after having eaten, or paediatric patients experiencing psychosomatic complaints (e.g. stomach ache).
  * For example, for the distraction module of the VR intervention, following paediatric patients can be recruited: paediatric patients undergoing a single medical (nursing procedure) such as (but not limited to) wound care, blood draw or vaccination.
* Age range of ≥ 4 and ≤ 16
* Normal or corrected-to-normal vision
* Normal or corrected-to-normal hearing

  * Note that in this study no specific medical procedure, treatment or patient population is chosen to increase the ecological validity of the study. In a real-life situation, the clinical staff chooses appropriate care methods (e.g. means of distraction or medication) based on their clinical expertise (in addition to treatment and pain management protocols). Therefore, the overall feasibility, acceptability, tolerability and initial clinical effect of the VR application are explored for an 'as-broad-as-possible' population, in order to provide information on what works best for whom with respect to Relaxation-VR. This practice-oriented approach allows us to investigate the potential of a VR intervention for a larger population, which could have the largest impact for the paediatric population and the clinical staff.

Exclusion Criteria:

* Patient has a history of seizure disorders (e.g. epilepsy)
* Physical impairment that preclude VR intervention (e.g. facial burns or wounds, contagious infectious disease, need for intensive care)
* Patient will undergo a medical procedure or treatment that is considered unsuitable in combination with the use of a VR headset, as assessed by the clinical staff (e.g., facial wound care)
* Non-Dutch native speaker: Both the paediatric patient and his/her caregiver must be able to provide informed consent and assent
* Previous enrolment in this study (during a previous hospital stay)

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Inpatient or outpatient in one of the study sites (UZ Brussel or AZ Sint-Maarten): each paediatric patient who will undergo a medical (nursing) procedure during the study period (1-01-2021 and 30-09-2021) and/or is in need of relaxation or distraction, as assessed by the clinical expertise of the involved clinical staff. Note that in this study no specific medical procedure, treatment or patient population is chosen to increase the ecological validity of the study.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-05-16 (Actual); Study Completion 2021-05-16 (Actual)

PRIMARY OUTCOMES:
Tolerability: Do participants experience symptoms of simulator sickness? (Pediatric Simulator Sickness Questionnaire) | Immediately after the intervention.
  This questionnaire is based on the Simulator Sickness Questionnaire (SSQ) and is used to assess physical adverse events due to the VR intervention. The query language of the SSQ was simplified for children and modified Wong-Baker faces were added to create a Peds SSQ, with a score of 0 (happy face) indicating no adverse event and a score of 6 (unhappy face) indicating more severe adverse event. The Peds SSQ, in accordance with the SSQ, contains queries that probe four symptom categories: eye strain, head and neck discomfort, sleepiness or fatigue, and dizziness or nausea. A lower score indicates a better outcome.
Feasibility as assessed by the paediatric participants | Immediately after the intervention
  Survey comprised of a combination of open-ended and response-set questions. Ease of use assessed with Visual Analogue Scale (VAS) ranging from 0 (very easy) to 100 (very difficult).
  Fun assessed with Visual Analogue Scale (VAS) ranging from 0 (A lot of fun to 100 (No fun at all).
Acceptability as assessed by the paediatric participants (Would you use it again? Would you recommend it to others?) | Immediately after the intervention
  Survey comprised of a combination of open-ended and response-set questions.
Feasibility as assessed by a parent of the paediatric patient | Immediately after the intervention
  Survey comprised of a combination of open-ended and response-set questions. E.g. Did the child keep the VR-headset on during the entire procedure?
Acceptability as assessed by a parent of the paediatric patient | Immediately after the intervention
  Survey comprised of a combination of open-ended and response-set questions. E.g., Why did you want to try it? Would you use it again?

SECONDARY OUTCOMES:
Changes in anxiety levels from pre-to-post intervention session: Visual Analogue Scale (VAS) | Immediately before and after the intervention.
  A visual analogue scale (VAS) for anxiety will be used to assess the anxiety levels. The VAS is a 10-cm horizontal line marked with the words "not anxious" (0, low score) at the left end and "very anxious" (100, high score) at the right end, with different facial expressions drawn along the line. The VAS is a widely used scale which is reliable and valid for measuring the subjective feelings of children.
Changes in pain levels from pre-to-post intervention session: Faces Pain Rating Scale-Revised (FPRS-R) | Immediately before and after the intervention.
  The FPS-R is a self-report measure used to assess the intensity of children's pain and comprises a scale of 0-10 comprising six horizontally arranged cartoon faces with expressions of "0 = no pain" to "10 = very painful". Participants will be asked to indicate the face that illustrates how much pain he/she feels. The FPS-R is shown to be appropriate for use in assessment of the intensity of children's acute pain from age 4 onward. The FPS-R is a reliable and valid scale for evaluating pain in children
Changes in emotion (happiness and arousal/stress) levels from pre-to-post intervention session: Two items of the Self-Assessment Manikin (SAM) | Immediately before and after the intervention.
  The Self-Assessment Manikin (SAM) is a non-verbal pictorial assessment technique that directly measures the pleasure, arousal, (and dominance = item that is left out) associated with a person's affective reaction to a wide variety of stimuli. A continuum of five stylized human figures (manikins) depicts feeling very happy (score of 1) to very sad (score of 9). For arousal, a second continuum of five stylized manikins depicts feeling very calm (score of 1) to very tense (score of 9). SAM is an inexpensive, easy method for quickly assessing reports of affective response in many contexts.

OTHER OUTCOMES:
Clinicians' assessment of usability: System Usability Scale (SUS) | Approximately after 16 weeks (After the last participant has finished the last session)
  Assessment of ease of use of the VR application with the System Usability Scale (SUS). The SUS is a 10-item questionnaire with five response options for respondents; from "strongly disagree" to "strongly agree" and returns scores ranging from 0 to 100. A higher SUS score indicates better usability.
Clinicians' satisfaction: Client Satisfaction Scale (CSQ-3) | Approximately after 16 weeks (After the last paediatric patient data is collected)
  Assessment of client satisfaction with the VR application with the Client Satisfaction Scale (CSQ-3). The CSQ-3 consists of 3 items with four response options and returns scores ranging from 8 to 32. Higher scores indicate higher satisfaction.
Clinicians' attitude towards Relaxation-VR via Unified Theory of Acceptance and Use of Technology (UTAUT) questionnaire | Approximately after 16 weeks (After the last paediatric patient data is collected)
  Assess clinicians' attitude towards technology with the Unified Theory of Acceptance and Use of Technology (UTAUT) questionnaire. The UTAUT questionnaire survey for end-users consists of 31 items with five response options ranging from "Totally disagree" (1) to "Totally agree" 5) and returns scores ranging from 31 to 155. The questionnaire survey consists of 7 subscales, for most of which higher scores indicate a more positive attitude towards the VR mirror therapy.
Exploration of barriers and facilitators of using VR in a hospital setting | Approximately after 16 weeks (After the last paediatric patient data is collected)
  Interview with clinicians.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - AZ Sint-Maarten, Mechelen, Antwerpen
  - UZ Brussel, Jette, Vlaams-Brabant

IPD SHARING:
Plan to Share IPD: No